CLINICAL TRIAL: NCT02508636
Title: Phase II Trial of Definitive Radiotherapy With Leuprolide and Enzalutamide in High Risk Prostate Cancer
Brief Title: Trial of Radiotherapy With Leuprolide and Enzalutamide in High Risk Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15558; NCI-2015-01757 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-08

CONDITIONS: Prostatic Neoplasms; Pelvic Nodal
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Leuprolide; Radiotherapy, Intensity-Modulated; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy: Enzalutamide, Leuprolide, Radiotherapy (Experimental): Participants will receive Enzalutamide: 160 mg per day, to begin within 0-7 days of the date of the first Luteinizing Hormone-Releasing Hormone (LHRH) agonist administration for total duration of 24 months as well as a single Leuprolide 7.5mg injection every month; single 22.5 mg injection every 3 months; single 30mg injection every 4 months; single 45 mg injection every 6-months based on the manufacturer for a total of 24 months.
  Radiation therapy should begin approximately 8 weeks (+/- 1 week) after the date of the first LHRH agonist/antagonist injection of hormone therapy is given and continue for a total of 5 weeks.
  Interventions: Drug: Enzalutamide; Drug: Leuprolide; Radiation: Intensity-Modulated Radiation Therapy

INTERVENTIONS:
Drug: Enzalutamide — Given orally
  Other Names: Xtandi
Drug: Leuprolide — Given via intramuscular injection
  Other Names: Lupron Depot
Radiation: Intensity-Modulated Radiation Therapy — A total dose of 45 Gy in 25 fractions of 1.8 Gy each.
  Other Names: Radiation Therapy; RT

SUMMARY:
This phase II trial studies the safety of giving enzalutamide with leuprolide acetate before and after radiation therapy and to see how well it works in treating patients with prostate cancer that is at high risk of returning. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Most types of prostate cancer also need testosterone to grow and spread. After radiation therapy, patients often receive treatments to reduce testosterone to prevent the cancer from returning. Leuprolide acetate works by reducing the amount of testosterone that the body makes. Enzalutamide is a stronger treatment that may block testosterone from reaching cancer cells. Adding enzalutamide to treatment with leuprolide acetate after radiation therapy may help prevent high-risk prostate cancer from returning and improve patient survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and safety of the combination of enzalutamide and leuprolide acetate (leuprolide) in patients undergoing definitive radiation therapy for high-risk prostate cancer or with pelvic nodal involvement.

II. To determine the prostate-specific antigen (PSA) complete response rate with the combination of enzalutamide and leuprolide (PSA-complete response (CR) as determined by PSA nadir =< 0.3) in patients undergoing radiation therapy for high-risk prostate cancer or pelvic nodal involvement.

SECONDARY OBJECTIVES:

I. To determine time to biochemical failure as determined by the American Society for Radiation Oncology (ASTRO) Phoenix definition of nadir + 2 ng/mL, local progression, regional progression, and distant metastases.

II. To determine time to clinical progression free survival III. To assess changes in PSA nadir and PSA and testosterone levels. IV. To assess changes in hemoglobin A1c (HbA1c), fasting glucose, fasting insulin and fasting lipid and cholesterol levels.

V. To document changes in quality of life outcomes.

EXPLORATORY OBJECTIVES:

I. To identify potential mutations and changes gene copy number associated with enzalutamide resistance in patients with high risk prostate cancer.

II. To identify gene expression patterns, splice variants, and gene signatures associated with enzalutamide treatment and enzalutamide resistance in patients with high risk prostate cancer.

III. To identify changes in the immune response with enzalutamide treatment.

OUTLINE:

Patients receive enzalutamide orally (PO) once daily (QD) and leuprolide acetate intramuscularly (IM) every 1, 3, 4, or 6 months for 24 months. Patients also undergo standard of care intensity-modulated radiation therapy (IMRT) 5 days per week for 5 weeks beginning at week 8, followed by optional brachytherapy. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6 weeks, 3-4 months, 6, 12, 18, 24, and 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of adenocarcinoma of the prostate within 180 days prior to registration at very high risk of recurrence as determined by 2 or more of the following combinations:

   * cT3a/b
   * PSA ≥20
   * Gleason score 8-10
   * ≥33% core involvement OR any patient with pelvic lymph node involvement ≥1cm as determined by pelvic CT or MRI imaging will meet eligibility criteria for enrollment.
2. Standard staging exams for patients with high-risk prostate cancer including bone scan or NaF Positron Emission Tomography (PET) /CT scan, and pelvic and prostate MRI.
3. No distant metastases (M0) on bone scan or NaF PET/CT within 90 days prior to registration. Equivocal bone scan findings are allowed if the physician determines that distant metastases are unlikely based on clinical judgment.
4. Zubrod Performance Status 0-2 within 60 days prior to enrollment.
5. Age ≥18
6. Complete blood count (CBC) with differential obtained within 30 days prior to registration on study, with adequate bone marrow function defined as follows:

   1. Absolute neutrophil count (ANC) ≥1,800 cells/mm3
   2. Platelets ≥100,000 cells/mm3
   3. Hemoglobin ≥8.0 g/dl (The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable)
   4. Serum creatinine <2.0 mg/dl and creatinine clearance >40 mL/min within 30 days prior to registration
   5. Bilirubin <1.5 x ULN and Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) <2 × ULN within 21 days prior to registration
7. Patients, even if surgically sterilized (i.e., status post vasectomy), who:

   1. Agree to practice effective barrier contraception during the entire study treatment period and for 4 months (120 days) after the last dose of study drug, or
   2. Agree to completely abstain from intercourse
8. Patient must be able to provide study-specific informed consent prior to study entry.

Exclusion Criteria:

1. Definite evidence of metastatic disease
2. Prior radical prostatectomy or bilateral orchiectomy for any reason
3. Prior invasive malignancy (except non-melanoma skin cancer) unless disease-free or not requiring systemic therapy for a minimum of 3 years.
4. Prior systemic chemotherapy for prostate cancer (Note that prior chemotherapy for a different cancer is allowed).
5. Prior radiotherapy, including brachytherapy, to the region of the prostate that would result in overlap of radiation therapy fields.
6. Previous hormonal therapy such as LHRH agonists (e.g. goserelin, leuprolide), anti-androgens (e.g. flutamide, bicalutamide), estrogens (e.g. DES), or surgical castration (orchiectomy)
7. Known hypersensitivity to enzalutamide or related compounds
8. History of adrenal insufficiency
9. Patients who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
10. Prior allergic reaction to the drugs involved in this protocol.
11. Cushing's syndrome
12. Severe chronic renal disease (serum creatinine >2.0 mg/dl and confirmed by creatinine clearance <40 mL/minute)
13. Chronic liver disease (bilirubin >1.5x ULN, ALT or AST >2x ULN)
14. Active/Uncontrolled Viral Hepatitis
15. Chronic treatment with glucocorticoids within one year.
16. History of seizure including febrile seizure or any condition that may predispose to seizure (e.g., prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization). Also, current or prior treatment with antiepileptic medications for the treatment of seizures or history of loss of consciousness or transient ischemic attack within 12 months prior to randomization.
17. Clinically significant cardiovascular disease including:

    1. Myocardial infarction within 6 months prior to screening
    2. Uncontrolled angina within 3 months prior to screening
    3. Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or subjects with history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multigated acquisition (MUGA) scan performed within 3 months results in a left ventricular ejection fraction that is ≥45%;
    4. History of clinically significant ventricular arrhythmias (e.g. ventricular tachycardia, ventricular fibrillation, torsades de pointes);
    5. History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
    6. Uncontrolled hypertension as indicated by a resting systolic blood pressure >170 mm Hg or diastolic blood pressure >105 mm Hg at screening. Patients with initially elevated systolic blood pressure >170 mm Hg or diastolic blood pressure >105 mm Hg are eligible if they undergo medical management and are re-screened.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hao Nguyen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Therapy: Enzalutamide and Leuprolide: Participants will receive Enzalutamide: 160 mg per day, to begin within 0-7 days of the date of the first Luteinizing Hormone-Releasing Hormone (LHRH) agonist administration for total duration of 24 months as well as a single Leuprolide 7.5mg injection every month; single 22.5 mg injection every 3 months; single 30mg injection every 4 months; single 45 mg injection every 6-months based on the manufacturer for a total of 24 months.
  Radiation therapy should begin approximately 8 weeks (+/- 1 week) after the date of the first LHRH agonist/antagonist injection of hormone therapy is given and continue for a total of 5 weeks.
Period: Overall Study
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 69.0 [50 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 11
Eastern Cooperative Oncology Group (ECOG) Scale of Performance Status [Number; unit: participants] — The ECOG Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themselves, their daily activity, and physical ability (walking, working, etc.). The scale/grade ranges from 0 to 5 with lower scores indicating a greater level of functioning.
  participants
    Score of 0 | 9
    Score of 1 | 2
    Score of 2 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Acute Treatment-related Toxicity
Description: Percentage of participants with acute, treatment-related toxicity defined as <=90 days within the completion of radiotherapy, for any treatment-related grade 3 or higher adverse events as classified by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: From start of treatment to 90 days after completion of radiotherapy, approximately 6 months total
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
percentage of participants | 36.36

2. Primary Outcome: Percentage of Participants With Late Treatment-related Toxicity
Description: Percentage of participants with late, treatment-related, toxicity is defined as any toxicity occurring >= 90 days from completion of radiotherapy for any grade 3 or higher treatment-related adverse events as classified by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: From 90 days after completion of radiotherapy until end of study, approximately 30 months total
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
percentage of participants | 27.27

3. Primary Outcome: Proportion of Patients Achieving a Prostate Specific Antigen-Complete Response (PSA-CR)
Description: A PSA measurement will be obtained at 120-127 days after initiation of androgen deprivation therapy. The proportion of patients achieving a PSA-CR (PSA nadir <=0.3) at 120-127 days will be determined.
Time Frame: Up to 127 days
Measure: Number; unit: proportion of participants
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
proportion of participants | 0.818

4. Secondary Outcome: Median Time to Biochemical Failure
Description: Prostate-specific antigen (PSA) nadir >=2 ng/mL, also known as the Phoenix definition, is the definition most commonly used to establish biochemical failure (BF) after external beam radiotherapy for prostate cancer management. Time to biochemical failure is defined as the time from start of treatment to the time of change in PSA >=2 ng/mL from the nadir.
Time Frame: Up to 36 months
Population: Only participants experiencing biochemical failure are reported
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 1
months | 36 [NA to NA] — Only 1 participant had biochemical failure at 36 months so there were not a sufficient number of events for a confidence interval to be computed

5. Secondary Outcome: Median Time to Local Failure
Description: Local failure was defined as the time from the start of treatment to a biopsy confirmed disease recurrence.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
months | NA [NA to NA] — No participants displayed local failure at 36 months so there were not a sufficient number of events for a confidence interval to be computed

6. Secondary Outcome: Number of Participants With Regional or Distant Metastases Over Time
Description: The number of participants with confirmed regional or distant metastases at 24 and 36 months will be reported.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
Participants
  Month 24 | 0
  Month 36 | 0

7. Secondary Outcome: Median Time to Clinical Progression
Description: Defined as the time from the start of study treatment to confirmed regional or distant metastases
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
months | NA [NA to NA] — No participants displayed clinical progression so there was an insufficient number of events to calculate median and confidence interval

8. Secondary Outcome: Overall Median Change in Hemoglobin A1c (HbA1c) Levels During Treatment
Description: HbA1C test results are reported as a percentage. The higher the percentage, the higher your blood sugar levels over the past two to three months. Changes in HbA1c results will be assessed during treatment and the overall median change in HbA1c will be reported.
Time Frame: Up to 24 months
Measure: Median (Full Range); unit: percentage
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
percentage | 0.2 [-1.1 to 1.5]

9. Secondary Outcome: Overall Median Change in Fasting Glucose Levels During Treatment
Description: Changes in fasting glucose levels results will be assessed during treatment and the overall median change in fasting glucose levels will be reported.
Time Frame: Up to 24 months
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
mg/dL | -2.7 [-20 to 19]

10. Secondary Outcome: Overall Median Change in Fasting Insulin Levels During Treatment
Description: Changes in fasting insulin levels will be assessed during treatment and the overall median change in fasting insulin levels will be reported.
Time Frame: Up to 24 months
Population: Data for fasting insulin was not collected
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 0

11. Secondary Outcome: Overall Median Change in Lipid Levels During Treatment
Description: Changes in fasting lipid levels will be assessed during treatment and the overall median change in fasting lipid levels will be reported.
Time Frame: Up to 24 months
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
mg/dL | 0 [-101 to 86]

12. Secondary Outcome: Overall Median Change in Total Cholesterol Levels During Treatment
Description: Changes in total cholesterol levels will be assessed during treatment and the overall median change in total cholesterol levels will be reported.
Time Frame: Up to 24 months
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
mg/dL | 12 [-270 to 86]

13. Secondary Outcome: Overall Median Change in High-Density Lipoprotein (HDL) Cholesterol Levels During Treatment
Description: Changes in fasting HDL levels will be assessed during treatment and the overall median change in fasting HDL will be reported.
Time Frame: Up to 24 months
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
mg/dL | 12 [-18 to 105]

14. Secondary Outcome: Overall Median Change in Low-Density Lipoprotein (LDL) Cholesterol Levels During Treatment
Description: Changes in fasting LDL levels will be assessed during treatment and the overall median change in fasting LDL will be reported.
Time Frame: Up to 24 months
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 11
mg/dL | 0 [-201 to 81]

15. Secondary Outcome: Overall Median Change in Score on the Expanded Prostate Cancer Index Composite (EPIC) During Treatment
Description: The Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment and assesses the disease-specific aspects of prostate cancer and its therapies and comprises four summary domains (Urinary, Bowel, Sexual and Hormonal). Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better health related quality of life. Changes in EPIC scores will be assessed during treatment and the overall median change in scores will be reported.
Time Frame: Up to 24 months
Population: Two participants did not complete the questionnaire
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 9
score on a scale
  Urinary incontinence | 6.25 [-20.8 to 25]
  Urinary Irritative/Obstructive | 6.25 [-6.25 to 25]
  Bowel | 0 [-20.8 to 4.2]
  Sexual | -44.4 [-56.9 to 0]
  Hormonal | -20 [-75 to 5]

16. Secondary Outcome: Overall Median Change in Patient-Reported Outcomes Measurement Information System (PROMIS) - Fatigue Scores During Treatment
Description: A PROMIS score of 50 is the average (or mean) score for a specific, relevant group of people under investigation. That group is the reference population. The PROMIS measures the responses use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. A score of 40 is one SD lower than the mean of the reference population and a score of 60 is one SD higher than the mean of the reference population. For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue). Changes in the PROMIS fatigue scores will be assessed during treatment and the overall median change in scores will be reported.
Time Frame: Up to 24 months
Population: Two participants did not complete the questionnaire
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 9
score on a scale | 0 [-9.6 to 21.5]

17. Secondary Outcome: Overall Median Change in EuroQol Group Five Dimensional Questionnaire (EQ-5D) During Treatment
Description: EQ-5D is a standardized instrument for measuring generic health status. The health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension by selecting one of the following responses: no problems (0), slight problems (1), mild problems (2), moderate problems (3), or severe problems (4) with a particular dimension. Lower scores indicate less issues/problems with that particular health dimension. Changes in the EQ-5D scores will be assessed during treatment and the overall median change in scores will be reported.
Time Frame: Up to 24 months
Population: Two participants did not complete the questionnaire
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 9
score on a scale
  Mobility | 0 [0 to 1]
  Self-Care | 0 [0 to 1]
  Usual Activities | 0 [0 to 1]
  Pain/Discomfort | 0 [0 to 2]
  Anxiety/Depression | 0 [0 to 1]

18. Secondary Outcome: Overall Median Change in EuroQol Group Visual Analog Scale (EQ-VAS) During Treatment
Description: The EQ-VAS records the patient's self-rated health on a vertical visual analogue scale, similar to a ruler, where the endpoints are labelled with 100='The best health you can imagine' on one end and 0='The worst health you can imagine' on the other, with 50 being the midpoint and participants mark an X on the scale to indicate how their health is on the day of the visit. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. Changes in the EQ-VAS scores will be assessed during treatment and the overall median change in scores will be reported.
Time Frame: Up to 24 months
Population: Two participants did not complete the questionnaire
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
Number analyzed (Participants) | 9
score on a scale | 72 [-2 to 81]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Groups:
- Combination Therapy: Enzalutamide and Leuprolide: Enzalutamide: 160 mg (for 40 mg capsules) per day; Oral administration to begin within 0-7 days of the date of the first Luteinizing Hormone-Releasing Hormone (LHRH) agonist administration for total duration of 24 months.
  Leuprolide: any duration formulation: single 7.5mg intramuscular injection every month; single 22.5 mg injection every 3 months; single 30mg injection every 4 months; single 45 mg injection every 6-months based on the manufacturer for a total of 24 months;
Arm/Group | Combination Therapy: Enzalutamide and Leuprolide
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy: Enzalutamide and Leuprolide (N=11)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy: Enzalutamide and Leuprolide (N=11)
Urinary frequency (Renal and urinary disorders) | 11 (40)
Urinary urgency (Renal and urinary disorders) | 10 (15)
Urinary retention (Renal and urinary disorders) | 4 (5)
Urinary incontinence (Renal and urinary disorders) | 3 (4)
Cystitis noninfective (Renal and urinary disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (2)
Hot flashes (Vascular disorders) | 11 (13)
Lymphedema (Vascular disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 9 (12)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Weight gain (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study closed earlier than expected which resulted in a low accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT02508636/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT02508636/ICF_001.pdf